CLINICAL TRIAL: NCT04067947
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending Single and Multiple Oral Dose Study of the Pharmacokinetics, Safety, and Tolerability of XG005 in Healthy Volunteers
Brief Title: Phase 1 Pharmacokinetics, Safety, and Tolerability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xgene Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: XG005-02
Record Dates: First submitted 2019-08-13; First posted 2019-08-28 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Investigator or designee, study coordinator(s), subjects, the Sponsor study team and its representatives, will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XG005 (Experimental): XG005 in 4 dose levels
  Interventions: Drug: XG005
- Placebo (Placebo Comparator): Placebo in all cohort
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: XG005 — XG005 Tablet
  Arms: XG005
Drug: Placebos — Placebo Tablet
  Arms: Placebo

SUMMARY:
A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending Single and Multiple Oral Dose Study of the Pharmacokinetics, Safety, and Tolerability of XG005 in Healthy Volunteers.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study which will investigate the PK, safety, and tolerability of four ascending single and multiple oral doses of XG005 in healthy subjects. The trial consists of two parts: a single ascending dose (SAD) PK evaluation (Part 1) and a multiple ascending dose (MAD) PK evaluation (Part 2). Approximately 32 Subjects will be enrolled sequentially into a total of 4 ascending dose levels in each part.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females between 18 and 55 years of age
2. BMI 18.0 to 30.0 kg/m2
3. Non-pregnant, non-breastfeeding female subjects

Exclusion Criteria:

1. Unstable or severe illness
2. History of, or current treatment for, GI disease
3. Clinically significant history of medical condition associated with GI events
4. History of or current glucose intolerance or gestational diabetes
5. Lifetime history of suicidal behavior
6. Creatinine clearance < 90 mL/min
7. Any elevation of liver function tests
8. Creatine kinase (CK) value of greater than 1.5 times the upper limit
9. Leucocytes or lymphocytes less than 1.5 times the lower limit of normal
10. Positive Hepatitis B surface antigen, HCV, or HIV

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Adverse Event related to XG005 | Day 1 to 7 days after last dose
  Adverse Event reported as mild, moderate, severe on physical exam, ECG and laboratory results

CONTACTS AND LOCATIONS:
Overall Officials: Feng Xu, PHD, Study Chair — Xgene Pharmaceutical Group
Locations (1):
- Linear Clinical Research Ltd, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No